CLINICAL TRIAL: NCT07060573
Title: Effects of Oral Stimulation Performed by Parents to Improve Sucking in Neonates Hospitalized in the NICU: A Randomized Clinical Trial
Brief Title: Effects of Oral Stimulation Performed by Parents to Improve Sucking in Neonates Hospitalized in the NICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Nelsi Alejandra Gonzalez Gonzalez, Physical Medicine and Rehabilitation Physician, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI 149/25
Record Dates: First submitted 2025-06-24; First posted 2025-07-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Premature Infant; Sucking Behavior
Keywords: Premature infant; sucking; oral stimulation; POFRAS; NICU; feeding; physiotherapy; Rehabilitation; parental involvement
MeSH Terms: conditions — Premature Birth; Sucking Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental Oral Stimulation Intervention (Experimental): Parents are trained to perform a standardized oral stimulation protocol (4 extraoral and 4 intraoral exercises) once daily for 14 days.
  Interventions: Behavioral: Parental Oral Stimulation Protocol
- Physiotherapist-led Oral Stimulation (Active Comparator): A licensed physiotherapist performs the same standardized oral stimulation protocol once daily for 14 days
  Interventions: Behavioral: Physiotherapist-led Oral Stimulation

INTERVENTIONS:
Behavioral: Parental Oral Stimulation Protocol — This intervention consists of a structured oral stimulation protocol composed of 4 extraoral and 4 intraoral exercises designed to improve oral motor function in preterm neonates. Exercises include perioral massage, stimulation of sucking reflex, and non-nutritive sucking using a pacifier. The protocol is administered once daily for 14 consecutive days. In this study arm, the intervention is performed by parents, previously trained and supervised in the neonatal unit.
  Arms: Parental Oral Stimulation Intervention
Behavioral: Physiotherapist-led Oral Stimulation — This intervention consists of a structured oral stimulation protocol composed of 4 extraoral and 4 intraoral exercises designed to improve oral motor function in preterm neonates. Exercises include perioral massage, stimulation of sucking reflex, and non-nutritive sucking using a pacifier. The protocol is administered once daily for 14 consecutive days. In this study arm, the intervention is performed by a licensed physiotherapist.
  Arms: Physiotherapist-led Oral Stimulation

SUMMARY:
This randomized clinical trial aims to evaluate the effectiveness of an oral stimulation program to improve sucking in preterm neonates hospitalized in the NICU. The study compares two groups: one receiving the intervention from a physiotherapist and the other from trained parents. The stimulation program includes 4 extraoral and 4 intraoral exercises applied once daily for 14 consecutive days. The primary outcome is improvement in the POFRAS score. Secondary outcomes include the time to exclusive oral feeding, nasogastric tube withdrawal, weight at discharge, hospital stay duration, and parental adherence. This study addresses the potential role of parent participation in neonatal rehabilitation in public hospitals with limited human resources.

DETAILED DESCRIPTION:
This single-blind, randomized clinical trial aims to compare the effectiveness of oral rehabilitation performed by trained parents versus physiotherapists to improve sucking in preterm neonates hospitalized in the NICU at the Hospital Civil de Guadalajara "Fray Antonio Alcalde," during the period July-October 2025.

Eligible neonates will be randomized into two groups:

Group A (Control): Intervention performed daily by a trained physiotherapist.

Group B (Experimental): Intervention performed daily by the parents after structured training and supervised implementation.

The oral stimulation program consists of 4 extraoral and 4 intraoral exercises designed to promote the development of sucking, swallowing, and breathing coordination. Each session lasts approximately 15 minutes and will be applied once daily for 14 consecutive days or until full oral feeding is achieved.

The primary outcome will be improvement in oral feeding readiness, assessed using the validated Spanish version of the POFRAS (Preterm Oral Feeding Readiness Assessment Scale). Secondary outcomes include: achievement of exclusive oral feeding, time to withdrawal of nasogastric tube, weight gain, hospital length of stay, and parent adherence to the protocol.

Randomization will use permuted blocks, and the outcome assessor will be blinded to group assignment. This study explores the feasibility and impact of parent-administered interventions in a public hospital setting with limited specialized personnel.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with corrected gestational age of 34 to 36 weeks
* Clinically stable to receive oral stimulation
* Informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Orofacial congenital malformations
* Severe neuromuscular disease
* Conditions contraindicating oral feeding

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in POFRAS Score from Day 1 to Day 14 | Baseline and Day 14 of intervention
  Change in the total score of the POFRAS scale (0-36 points), which evaluates oral feeding readiness in preterm neonates. A higher score indicates greater readiness for oral feeding.

SECONDARY OUTCOMES:
Time to Exclusive Oral Feeding | From baseline to achievement of full oral feeding (up to 14 days)
  Number of days required for the neonate to transition from tube feeding to exclusive oral feeding without need for nasogastric support.
Weight at Hospital Discharge | Baseline and Day 14 post-intervention
  Body weight in grams recorded at the time of NICU discharge
Length of Hospital Stay | From birth until hospital discharge, assessed up to 60 days
  Total number of days the neonate remains hospitalized in the neonatal intensive care unit (NICU) until medically cleared for discharge.
Parental Satisfaction | At Day 14 or end of intervention
  Level of parental satisfaction with the intervention protocol, assessed using a 5-point Likert scale (1 = very dissatisfied; 5 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Antiguo Hospital Civil Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) due to institutional data privacy policies and the absence of a secure data-sharing infrastructure. Data will remain confidential and stored locally, in compliance with ethical and regulatory standards.